CLINICAL TRIAL: NCT04718116
Title: Management of Postsurgical Pain After Cardiac Operations: Comparison of Tapentadol and Tramadol Analgesia
Brief Title: Tapentadol Versus Tramadol Analgesia Post Cardiac Surgery
Acronym: vasso-annie
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 668/24.02.2020
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain; Surgery; Pain, Postoperative; Pain, Acute; Pain, Chronic; Pain, Procedural; Pain, Neuropathic; Analgesia
Keywords: tapentadol; tramadol
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Pain, Procedural; Neuralgia; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tapentadol 50 mg (Active Comparator): tapentadol 50mg p.o 3 times daily for two days
  Interventions: Drug: Group tapentadol 50 mg
- tapentadol 75 mg (Active Comparator): tapentadol 75 mg p.o 3 times daily for two days
  Interventions: Drug: group tapentadol 75 mg
- tramadol 100 mg (Active Comparator): tramadol 100 mg p.o 3 times daily for two days
  Interventions: Drug: group tramadol 100 mg

INTERVENTIONS:
Drug: Group tapentadol 50 mg — patients in group A will receive tapentadol 50 mg p.o 3 times daily for two days
  Other Names: group A
  Arms: tapentadol 50 mg
Drug: group tapentadol 75 mg — patients in group B will receive tapentadol 75 mg p.o 3 times daily for two days
  Other Names: group B
  Arms: tapentadol 75 mg
Drug: group tramadol 100 mg — patients in group C will receive tramadol 100 mg p.o 3 times daily for two days
  Other Names: group C
  Arms: tramadol 100 mg

SUMMARY:
The aim of this randomized one-blinded study will be to evaluate the efficacy and tolerability of two different oral doses of tapentadol and compare it to tramadol (an opioid commonly used to treat post-surgical pain) in cardiac surgery patients

DETAILED DESCRIPTION:
Management of post-surgical pain is a daily challenge for every anaesthetist. Undertreated post-surgical pain can result in cardiovascular, pulmonary and gastrointestinal complications, as well as chronic pain and negative psychological effects. A negative impact may be seen on immune function, coagulation and wound healing. Opioids have been the cornerstone in the treatment of pain after cardiac surgery. However, opioids have a number of adverse effects such as respiratory depression, gastrointestinal alterations, dizziness, delirium, addiction.

Tapentadol is a new synthetic opioid with dual mechanism of action. It acts as a mu-receptor agonist, as well as norepinephrine reuptake inhibitor. It is used to treat moderate to severe pain and is associated with fewer adverse effects compared to other opioids.

The aim of this randomized one-blinded study will be to evaluate the efficacy and tolerability of two different oral doses of tapentadol and compare it to tramadol (an opioid commonly used to treat post-surgical pain).

Patients undergoing cardiac surgery and being discharged from ICU to ward within 30 hours of surgery, will be divided into 3 groups. Group A will receive tapentadol 50mg p.o 3 times daily for two days, group B will receive tapentadol 75 mg p.o 3 times daily for two days and group C will receive tramadol 100 mg p.o 3 times daily for two days. Pain level will be assessed with Numeric Rating Scale (NRS), before drug administration and two hours after drug administration. Overall patient satisfaction will be assessed with Likert scale. Brief Pain Inventory( short form) and DN4 questionnaire will be used to detect chronic pain and neuropathic pain respectively, 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age <75 years old
* patients discharged from Intensive Care Unit (ICU) in less than 30 hours
* elective cardiac surgery

Exclusion Criteria:

* hepatic failure (increased transaminase levels
* renal failure (creatinine> 2 mg/dL)
* ileus
* emergency surgery (hemorrhage, tamponade, aortic dissection)
* readmission in ICU
* treatment with monoaminoxidase inhibitors, selective serotonine reuptake inhibitors or antiepileptics
* age>75 years old
* communication or language barriers
* Lack of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline in pain score at rest | 2 hours after analgesia administration
  pain score will be assessed by the use of Numeric Rating Scale (NRS) 2 hours after analgesia administration, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
change from baseline in pain score during coughing | 2 hours after analgesia administration
  pain score will be assessed by the use of Numeric Rating Scale (NRS) 2 hours after analgesia administration, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
side effects | 2 hours after analgesia administration
  side effects resulting from analgesic administration, yes or no
incidence of chronic pain 3 months after surgery | 3 months after surgery
  occurrence of chronic pain at the site of the operation 3 months after surgery, with the use of the Brief Pain Inventory Questionnaire
incidence of chronic pain 6 months after surgery | 6 months after surgery
  occurrence of chronic pain at the site of the operation 6 months after surgery, with the use of the Brief Pain Inventory Questionnaire
incidence of neuropathic pain 3 months after surgery | 3 months after surgery
  occurrence of neuropathic pain 3 months after surgery, with the use of the Douleur Neuropathique (DN4) Questionnaire
incidence of neuropathic pain 6 months after surgery | 6 months after surgery
  occurrence of neuropathic pain 6 months after surgery, with the use of the Douleur Neuropathique (DN4) Questionnaire

SECONDARY OUTCOMES:
hospitalization time | postoperatively, an average period of 10 days
  duration of hospital stay after surgery in days
satisfaction from postoperative analgesia | 72 hours postoperatively
  satisfaction from postoperative analgesia on a six-point Likert scale with 1 marked as minimal satisfaction and 6 as maximal satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (2):
- Greece (2):
  - Onassis Cardiac Surgery Centre, Athens
  - Ygeia General Hospital of Athens, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raksamani K, Wongkornrat W, Siriboon P, Pantisawat N. Pain management after cardiac surgery: are we underestimating post sternotomy pain? J Med Assoc Thai. 2013 Jul;96(7):824-8. PMID 24319854
- [Background] Roediger L, Larbuisson R, Lamy M. New approaches and old controversies to postoperative pain control following cardiac surgery. Eur J Anaesthesiol. 2006 Jul;23(7):539-50. doi: 10.1017/S0265021506000548. PMID 16677435
- [Background] Taillefer MC, Carrier M, Belisle S, Levesque S, Lanctot H, Boisvert AM, Choiniere M. Prevalence, characteristics, and predictors of chronic nonanginal postoperative pain after a cardiac operation: a cross-sectional study. J Thorac Cardiovasc Surg. 2006 Jun;131(6):1274-80. doi: 10.1016/j.jtcvs.2006.02.001. PMID 16733157
- [Background] Gjeilo KH, Klepstad P, Wahba A, Lydersen S, Stenseth R. Chronic pain after cardiac surgery: a prospective study. Acta Anaesthesiol Scand. 2010 Jan;54(1):70-8. doi: 10.1111/j.1399-6576.2009.02097.x. Epub 2009 Aug 13. PMID 19681771
- [Background] Nachiyunde B, Lam L. The efficacy of different modes of analgesia in postoperative pain management and early mobilization in postoperative cardiac surgical patients: A systematic review. Ann Card Anaesth. 2018 Oct-Dec;21(4):363-370. doi: 10.4103/aca.ACA_186_17. PMID 30333328
- [Background] Tzschentke TM, Christoph T, Kogel BY. The mu-opioid receptor agonist/noradrenaline reuptake inhibition (MOR-NRI) concept in analgesia: the case of tapentadol. CNS Drugs. 2014 Apr;28(4):319-29. doi: 10.1007/s40263-014-0151-9. PMID 24578192
- [Background] Langford RM, Knaggs R, Farquhar-Smith P, Dickenson AH. Is tapentadol different from classical opioids? A review of the evidence. Br J Pain. 2016 Nov;10(4):217-221. doi: 10.1177/2049463716657363. Epub 2016 Jul 25. PMID 27867511
- [Background] Raffa RB, Buschmann H, Christoph T, Eichenbaum G, Englberger W, Flores CM, Hertrampf T, Kogel B, Schiene K, Strassburger W, Terlinden R, Tzschentke TM. Mechanistic and functional differentiation of tapentadol and tramadol. Expert Opin Pharmacother. 2012 Jul;13(10):1437-49. doi: 10.1517/14656566.2012.696097. Epub 2012 Jun 15. PMID 22698264
- [Background] Lee YK, Ko JS, Rhim HY, Lee EJ, Karcher K, Li H, Shapiro D, Lee HS. Acute postoperative pain relief with immediate-release tapentadol: randomized, double-blind, placebo-controlled study conducted in South Korea. Curr Med Res Opin. 2014 Dec;30(12):2561-70. doi: 10.1185/03007995.2014.954665. Epub 2014 Aug 27. PMID 25133962